CLINICAL TRIAL: NCT04371978
Title: Efficacy and Safety of Dipeptidyl Peptidase-4 Inhibitors in Diabetic Patients With Established COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: End of COVID-19 outbreak in Israel
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Ran Abuhasira, Dr. Ran Abuhasira, Internal Medicine B, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0303-20-RMC
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: COVID 19; Coronavirus; Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases; Dipeptidyl-Peptidase IV Inhibitors; Linagliptin; Severe Acute Respiratory Syndrome Coronavirus 2; Sars-CoV2; Hypoglycemic Agents; Respiratory Tract Diseases; Incretins; Hormones
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Diabetes Mellitus, Type 2; Diabetes Mellitus; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Respiratory Tract Diseases | interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPP-4 inhibition (Experimental): Participants in the Dipeptidyl Peptidase-4 (DPP-4) inhibition group will receive linagliptin in addition to standard of care insulin regimen as per hospital protocol during their entire hospitalization.
  Interventions: Drug: Linagliptin 5 MG
- Control (No Intervention): Participants in the control group will receive only the standard of care insulin regimen as per hospital protocol during their entire hospitalization.

INTERVENTIONS:
Drug: Linagliptin 5 MG — Linagliptin 5 mg PO once daily
  Other Names: Trajenta
  Arms: DPP-4 inhibition

SUMMARY:
The coronavirus disease 2019 (COVID-19) is an emerging pandemic in 2020 caused by a novel coronavirus named SARS-CoV2. Diabetes confers a significant additional risk for COVID-19 patients. Dipeptidyl peptidase 4 (DPP-4) is a transmembrane glycoprotein expressed ubiquitously in many tissues. In addition to its effect on glucose levels, DPP-4 has various effects on the immune system and several diseases, including lung diseases. This trial aims to assess the safety and efficacy of linagliptin, a DPP-4 inhibitor, in the treatment of COVID-19. The trial will be randomized without blinding, with one are treated by insulin only for glucose balance and the other by insulin and linagliptin. The trial will assess the effects of linagliptin on different measures of COVID-19 recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. History of or type 2 diabetes mellitus or a diagnosis of type 2 diabetes during hospitalization.
3. Confirmation of infection with SARS-CoV-2 by PCR testing.
4. Patients within 10 days from symptom onset or patients within 48 hours after laboratory diagnosis (SARS-CoV-2 PCR).

Exclusion Criteria:

1. WHO COVID-19 Ordinal Scale for Clinical Improvement ≥ 6.
2. Respiratory failure requiring mechanical ventilation prior to randomization.
3. Use of vasopressor or inotropic medications prior to randomization.
4. Intolerance/hypersensitivity to dipeptidyl peptidase-4 inhibitors.
5. Patients expected to require intensive care unit admission or immediate surgical intervention.
6. Participation in another trial assessing any treatment for COVID-19.
7. Current treatment with a DPP-4 inhibitor.
8. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Time to clinical change | 28 days
  Clinical change is defined as 2 points reduction in the World Health Organization (WHO) Ordinal Scale for Clinical Improvement of COVID-19: 0 - No clinical or virological evidence of infection; 1 - No limitation of activities; 2 - Limitation of activities; 3 - Hospitalized, no oxygen therapy; 4 - Oxygen by mask or nasal prongs; 5 - Non-invasive ventilation or high-flow oxygen; 6 - Intubation and mechanical ventilation; 7 - Ventilation + additional organ support - pressors, renal replacement therapy, extracorporeal membrane oxygenation; 8 - Death.

SECONDARY OUTCOMES:
Percent of serious adverse events and premature discontinuation of treatment. | 28 days
Percent of patients with clinical improvement. | 28 days
  Percent of patients with a 2 points reduction in the World Health Organization (WHO) Ordinal Scale for Clinical Improvement of COVID-19.
Length of hospitalization. | 28 days
All-cause mortality. | 28 days
Percent of supplemental oxygen use. | 28 days
Supplemental oxygen-free days. | 28 days
Percent of mechanical ventilation use. | 28 days
Ventilator-free days. | 28 days
Percent of ICU admissions. | 28 days
ICU-free days. | 28 days
Percent of 50% decrease in C-reactive protein (CRP) levels | Up to 28 days
Time to virologic response, defined as no detection of SARS-CoV-2 in a PCR test. | 28 days

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Rabin Medical Center, Hasharon Campus, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abuhasira R, Ayalon-Dangur I, Zaslavsky N, Koren R, Keller M, Dicker D, Grossman A. A Randomized Clinical Trial of Linagliptin vs. Standard of Care in Patients Hospitalized With Diabetes and COVID-19. Front Endocrinol (Lausanne). 2021 Dec 22;12:794382. doi: 10.3389/fendo.2021.794382. eCollection 2021. PMID 35002970